CLINICAL TRIAL: NCT01166009
Title: Protocol For A Research Database For Hematopoietic Stem Cell Transplantation, Other Cellular Therapies and Marrow Toxic Injuries
Brief Title: CIBMTR Research Database
Status: Recruiting | Type: Observational
Sponsor: Center for International Blood and Marrow Transplant Research (Network)
Responsible Party: Sponsor
Other Study IDs: NMDP IRB-2002-0063; NCT00923585 (obsolete NCT alias); NCT01160497 (obsolete NCT alias); NCT02401009 (obsolete NCT alias)
Record Dates: First submitted 2010-07-16; First posted 2010-07-20 (Estimated); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Autologous Stem Cell Transplantation; Allogeneic Stem Cell Transplantation; Solid Tumors; Blood Cancers; CAR-T; Gene Therapy; Non-malignant Disease
Keywords: Data Collection; CIBMTR; NMDP; Stem Cell Transplantation; Gene Therapy; CAR-T
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
The primary purpose of the Research Database is to have a comprehensive source of observational data that can be used to study HSC transplantation and cellular therapies.

A secondary purpose of the Research Database is to have a comprehensive source of data to study marrow toxic injuries.

Objectives:

To learn more about what makes stem cell transplants and cellular therapies work well such as:

* Determine how well recipients recover from their transplants or cellular therapy;
* Determine how recovery after a transplant or cellular therapy can be improved;
* Determine how a donor's or recipient's genetics impact recipient recovery after a transplant or cellular therapy;
* Determine how access to transplant or cellular therapy for different groups of patients can be improved;
* Determine how well donors recover from the collection procedures.

ELIGIBILITY:
Eligibility to Participate in the Research Database

Recipient Eligibility Criteria:

* Any recipient of an unrelated or related donor or autologous HSC transplant in a CIBMTR center is eligible to participate in the Research Database. This includes adults with and without decision making capacity, and children.

Individual with Marrow Toxic Injury Eligibility Criteria:

* Any individual who is treated for a marrow toxic injury at a center participating in the NMDP's Radiation Injury Transplant Network (RITN) is eligible to participate in the Research Database. This includes adults with and without decision making capacity, and children. Eligible individuals may have received supportive care only, growth factor support, HSC transplant or other appropriate medical treatment for marrow toxic injury. Treatments applied are at the discretion of the care facility, and are not determined by the NMDP or CIBMTR.

Unrelated Donor Eligibility Criteria:

* All donors registered on the NMDP Registry who have been requested to donate a product for a recipient are eligible to participate in the Research Database.
* All maternal cord blood donors are enrolled in the NMDP Cord Blood Bank Investigational New Drug (IND) protocol, and sign an informed consent document specific to that protocol. Data collected as part of the Cord Blood Bank protocol are included in the Research Database.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Recipients and Donors that are involved with stem cell transplantation, other cellular therapies, and gene therapies.
Sampling Method: Non-Probability Sample
Enrollment: 99999999 (Estimated)
Dates: Start 2002-07; Primary Completion 2050-07 (Estimated); Study Completion 2050-07 (Estimated)

PRIMARY OUTCOMES:
A Comprehensive Source of Observational Data to assess Stem Cell Transplant | Anually - on average
  A primary outcome is to have a comprehensive source of stem cell transplant data that can be used to assess topics such as:
  * Recipient Recover time
  * How recovery after transplant and other cellular therapies can be improved
  * Long term outcomes after transplantation and other cellular therapies
  * How well donors recover from collection procedure

SECONDARY OUTCOMES:
A Comprehensive Source of Data for Marrow Toxic Injuries | anually- on average
  In the event of a radiation exposure accident, the NMDP has a radiation injury treatment network, whose purpose is to collect data to understand the outcomes of patients treated under these circumstances. Any patient who is treated for a marrow toxic injury at a center participating in the NMDP's Radiation Injury Treatment Network (RITN) is eligible to participate in the Research Database.
Prospective Assessment of Allogeneic Hematopoietic Cell Transplantation in Patients with Medicare Coverage (17-CMS-SCD) | annually - on average
  This protocol supports data collection for a sub study titled 17-CMS-SCD, an observational study to compare survival of patients 15 to 50 years of age with sickle cell disease who receive allogeneic transplantation compared to those receiving standard of care treatments.
  * To provide a mechanism to Medicare Beneficiaries with sickle cell disease for claims coverage for allogenic hematopoietic cell transplant.
  * To provide data requested by Medicare under its coverage with evidence development (CED) process to make payment on claims for HCT using the existing research observational database for the CIBMTR
Prospective Assessment of Allogeneic Hematopoietic Cell Transplantation in Patients with Medicare Coverage (10CMSMDS-1) | annually - on average
  This protocol supports data collection for a sub-study titled 10-CMSMDS-1 with objective to prospectively examine outcomes of allogenic hematopoietic cell transplant in adults >= 65 years of age with myelodysplastic syndrome to determine whether their outcomes are similar to those in younger patients.
  * To provide a mechanism for Medicare Beneficiaries with myelodysplastic syndrome for claims coverage for allogenic hematopoietic cell transplant
  * To provide data requested by Medicare under its CED to make payment on claims for HCT using the existing research observational database of the CIBMTR"

OTHER OUTCOMES:
Prospective Assessment of Allogeneic Hematopoietic Cell Transplantation in Patients with Medicare Coverage | annually - on average
  This study is the main protocol for the following two sub studies. Details for these sub-studies are found under separate NCT numbers.
  * Multiple Myeloma Medicare Study (NCT03127761): 17-CMS-MM
  * Myelofibrosis Medicare Study (NCT02934477): 16-CMS-MF

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Steinert, PhD, MBA, Principal Investigator — Center for International Blood and Marrow Transplant Research
Locations (2):
- United States (2):
  - Center for International Blood and Marrow Transplant Research, Minneapolis, Minnesota
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Atallah E, Logan B, Chen M, Cutler C, Deeg J, Jacoby M, Champlin R, Nishihori T, Confer D, Gajewski J, Farnia S, Greenberg P, Warlick E, Weisdorf D, Saber W, Horowitz MM, Rizzo JD. Comparison of Patient Age Groups in Transplantation for Myelodysplastic Syndrome: The Medicare Coverage With Evidence Development Study. JAMA Oncol. 2020 Apr 1;6(4):486-493. doi: 10.1001/jamaoncol.2019.5140. PMID 31830234